CLINICAL TRIAL: NCT06388148
Title: Efficacy and Safety of Endovascular Thrombectomy Plus Medical Management Versus Medical Management Alone in Acute Ischemic Stroke Patients With Large Vessel Occlusion and Extra-Large Infarct Core: A Multicenter, Randomized Controlled Trial
Brief Title: Endovascular Treatment for eXtra-Large Ischemic Stroke
Acronym: XL STROKE-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongming Qiu (Other)
Collaborators: The First Affiliated Hospital, University of South China (Unknown); Xiangtan Central Hospital (Other); Affiliated Hangzhou First People's Hospital, School of Medicine, Westlake University (Unknown); Longyan First Affiliated Hospital of Fujian Medical University (Unknown); Taizhou First People's Hospital (Other); Zhangzhou Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor-Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Organization: Xinqiao Hospital of Chongqing (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XL STROKE-2
Record Dates: First submitted 2024-04-21; First posted 2024-04-29 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Stroke, Acute Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Practice Management, Medical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular thrombectomy (Experimental): Patients in this group will be treated with medical management plus endovascular thrombectomy
  Interventions: Drug: Medical management; Procedure: Endovascular thrombectomy
- Medical management (Active Comparator): Patients in this group will be treated with medical management alone
  Interventions: Drug: Medical management

INTERVENTIONS:
Drug: Medical management — Medical management includes IV thrombolysis, antiplatelet, and/or anticoagulation.
Procedure: Endovascular thrombectomy — Endovascular thrombectomy with stent-retriever, local aspiration, angioplasty, and/or stenting.
  Arms: Endovascular thrombectomy

SUMMARY:
The role of endovascular thrombectomy in patients with extra-large ischemic burden is still unclear. The XL STROKE-2 randomized trial is aiming to investigate the efficacy and safety of mechanical thrombectomy in acute extra-large ischemic stroke patients with large vessel occlusion.

DETAILED DESCRIPTION:
Several randomized trials have shown that endovascular thrombectomy improve functional outcomes in acute ischemic stroke patients with large vessel occlusion. Recently, six randomized controlled trials demonstrated the efficacy and safety of endovascular thrombectomy for large infarct patients (defined as Alberta Stroke Program Early Computed Tomography Score [ASPECTS] ≥3 or infarct core <100ml). Patients with extra-large infarct core (volume greater than 100 mL, ASPECTS score of 0 to 2) accounted for a small proportion of these trials. Therefore, the role of endovascular thrombectomy in patients with extra-large ischemic burden is still unclear. That is to say, exactly where the lower limit of endovascular thrombectomy is unknown. The XL STROKE-2 randomized trial is aiming to investigate the efficacy and safety of mechanical thrombectomy in acute extra-large ischemic stroke patients with large vessel occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, and modified Rankin scale score = 0 or 1 in patients 80 years or older;
2. Acute ischemic stroke within 6 hours from last known well to randomization, or with negative MRI-FLAIR (no change on FLAIR sequence and presence of infarct on MRI-DWI) if > 6 hours or unknown last known well time;
3. Occlusion of the internal carotid artery, M1 or M2 segment of the middle cerebral artery confirmed by CTA/MRA/DSA;
4. Baseline ASPECTS score of 0-2 or infarct core volume ≥100ml;
5. The patient or patient's representative signs a written informed consent form.

Exclusion Criteria:

1. CT or MR evidence of hemorrhage;
2. Evidence of mass effect with ventricular effacement, midline shift or herniation on baseline imaging;
3. Vessel tortuosity where it is expected that the thrombectomy device will not be able to reach the occlusion site or result in unstable access;
4. History of bleeding disorders, severe heart, liver or kidney disease, or sepsis;
5. Currently participating in another investigational drug study;
6. Any terminal illness with life expectancy less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2024-06-16 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale score | 90 days after randomization
  Modified Rankin scale score (mRS): scores range from 0 to 6, with 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death

SECONDARY OUTCOMES:
Rate of successful reperfusion | Within 5 minutes at the end of angiogram
  Final reperfusion grade of 2b-3 on eTICI scale (This 7-point compilation of TICI grades, termed the expanded TICI (eTICI), reflects all previously reported thresholds used to define reperfusion after endovascular stroke therapy. In brief, eTICI grade 0 is equivalent to no reperfusion or 0% filling of the downstream territory; eTICI 1 reflects thrombus reduction without any reperfusion of distal arteries; eTICI 2a is reperfusion in less than half or 1-49% of the territory; eTICI 2b50 is 50-66% reperfusion, exceeding the modified TICI (mTICI) 2B threshold but below the original TICI 2B cut-off point; eTICI 2b67 is 67-89% reperfusion, exceeding TICI but below TICI 2C; eTICI 2c is equivalent to TICI 2C or 90-99% reperfusion; and eTICI 3 is complete or 100% reperfusion, tantamount to TICI 3.)
Rate of excellent outcome | 90 days after randomization
  Score of 0-1 on the modified Rankin scale
Rate of functional independence | 90 days after randomization
  Score of 0-2 on the modified Rankin scale
Rate of independent ambulation | 90 days after randomization
  Score of 0-3 on the modified Rankin scale

CONTACTS AND LOCATIONS:
Overall Officials: Guangxiong Yuan, Principal Investigator — Xiangtan Central Hospital; Congguo Yin, Principal Investigator — Hangzhou First Hospital of Zhejiang University; Tingyu Yi, Principal Investigator — Zhangzhou Affiliated Hospital of Fujian Medical University; Chong Zheng, Principal Investigator — Longyan First Hospital of Fujian Medical University; Chenghua Xu, Principal Investigator — Taizhou First People's Hospital; Zhongfan Ruan, Principal Investigator — The First Affiliated Hospital, Hengyang Medical School, University of South China
Locations (2):
- China (2):
  - The First Affiliated Hospital, Hengyang Medical School, University of South China, Hengyang, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Two years after the trial results are revealed.
Access Criteria: After approval of a proposal from principal investigator